CLINICAL TRIAL: NCT07333430
Title: A Phase 1a/1b Open-Label Study With Dose Escalation and Expansion Phases to Evaluate Safety and Preliminary Efficacy of Naïve HBI0101 CART Therapy for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Naive HBI0101 CAR-T Therapy in Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Polina Stepensky, Prof. Polina Stepensky, Director Department of Bone Marrow Transplantation and Cancer Immunotherapy, Hadassah Medical Organization, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Naive HBI0101-1 CAR-T
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Multiple Myeloma (MM)
Keywords: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Naïve BCMA (Experimental): The dose escalation phase (Part 1a) will follow a 3+3 design and include up to 3 dose level cohorts. Eligible participants for Cohorts 1, 2, and 3 will receive a single (low, medium or high) dose of 80 × 106 ± 30%, 160 × 106 ± 25% and 240 × 106 ± 20% Naïve HBI0101 CART.
  The expansion phase (Part 1b) will receive up to Maximum Tolerated Dose (MTD) .
  Interventions: Biological: Naive HBI0101 CAR-T

INTERVENTIONS:
Biological: Naive HBI0101 CAR-T — Naïve HBI0101 CART is defined as autologous T cells transduced ex-vivo with anti-BCMA CAR retroviral vector encoding the chimeric antigen receptor (CAR) targeted to human BCMA. The Naïve HBI0101 CART is provided cryopreserved.

SUMMARY:
A Phase 1a/1b Open-Label Study with Dose Escalation and Expansion Phases to Evaluate Safety and Preliminary Efficacy of Naïve HBI0101 CART Therapy for the Treatment of Relapsed/Refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age at the time of signing informed consent.
2. Voluntarily signed informed consent form.
3. Diagnosis of relapsed/refractory multiple myeloma (Parts 1a and 1b), with measurable disease at screening visit as follows:

   Multiple Myeloma (at least one of the criteria below):
   1. Serum M-protein greater or equal to 0.5 g/dL.
   2. Urine M-protein greater or equal to 200 mg/24 h.
   3. Serum free light chain (FLC) assay: involved FLC level greater or equal to 3 mg/dL (30 mg/L) provided serum FLC ratio is abnormal.
   4. A biopsy-proven evaluable plasmacytoma*.
   5. Bone marrow plasma cells > 10% of total bone marrow cells*.
   6. Non secretory patient will be allowed provided they have measurable disease by PET-CT or bone marrow aspiration, as designated*.

      * Results pre-dating the Screening visit by up to 28 days may be used to establish eligibility.
4. R/R MM subjects must have been exposed to at least three prior lines of therapy including the following agents:

   1. proteasome inhibitor
   2. immunomodulatory (IMiDs) agent
   3. anti-CD38 antibody
5. For part 1a: At least one of the following risk factors: a. Extra-medullary disease (EMD) - defined as a MM lesion that is not connected to a bone. b. previous exposure to an anti-BCMA therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
7. Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.
8. Recovery to ≤ Grade 2 or baseline of any non-hematologic toxicities due to prior treatments, excluding alopecia and Grade 3 neuropathy, and toxicities that are irreversible and not expected to interfere with study treatment or pose safety concerns, per investigator judgement.
9. Ability and willingness to adhere to the study visit schedule and all protocol requirements.
10. For subjects with relapsed multiple myeloma who have previously undergone allogenic stem cell transplantation: no evidence of graft versus host disease after cessation of any immunosuppressive therapy for at least one month before recruitment to the study.

Exclusion Criteria:

1. Contraindication to a study treatment/procedure or is anticipated to receive treatment/procedure that may preclude performance of study procedures.
2. Known bulky central nervous system disease.
3. Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) and/or direct bilirubin > 4x ULN.
4. Inadequate renal function defined by estimated clearance of <20(ml/min).
5. International ratio (INR) or partial thromboplastin time (PTT) > 2 x ULN, unless on a stable dose of anticoagulant for a thromboembolic event (provided this event is not an exclusion criteria).
6. Inadequate bone marrow function defined by absolute neutrophil count (ANC) < 1000 cells/mm3, platelet count < 30,000 mm3, or hemoglobin < 8 g/dL. Subjects with absolute lymphocyte count < 300 cells/mm3 may be excluded (due to potential challenges with producing CART), per investigator judgement.
7. Left ventricular ejection fraction < 40%.
8. Ongoing treatment with chronic immunosuppressant such as cyclosporine or systemic steroids (physiological replacement doses of steroids are allowed up to 12 mg/m2/d hydrocortisone or equivalent)
9. Significant co-morbid condition or disease which in the judgment of the Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, recent significant traumatic injury, and other conditions.
10. Known human immunodeficiency virus (HIV) positive status.
11. Active Hepatitis B active infection (defined as HBS-antigen and HBV DNA positive) or Hepatitis C active infection (defined as anti-HCV and HCV RNA positive).
12. Active CMV infection.
13. Known history of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within 3 months.
14. Chronic atrial fibrillation with uncontrolled heart rate.
15. Second primary malignancy that has required therapy in the last 2 years or is not in complete remission. This exclusion criterion does not exclude the following subjects: successfully treated non- metastatic basal cell or squamous cell skin carcinoma, or prostate cancer under control with hormonal therapy
16. Subjects who have had a venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation and who meet any of the following criteria:

    1. Have been on a stable dose of anticoagulation for < 1 month (except for acute line insertion induced thrombosis.
    2. Have had a Grade 2, 3, or 4 hemorrhage in the last 30 days
    3. Are experiencing continued symptoms from their venous thromboembolic event (e.g. continued dyspnea or oxygen requirement).
17. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the Maximum Tolerated Dose (MTD) | 21 days after infusion
  MTD will be determined by dose limiting toxicities
Evaluate safety of Naïve HBI0101 CART in Parts 1a and 1b | 24 Months after infusion
  Incidence of Serious Adverse Events and Adverse Events of Special Interest related to study treatment.

SECONDARY OUTCOMES:
Evaluate clinical response to Naïve HBI0101 CART | 24 Months after infusion
  Overall response rate- Percentage of participants who achieved at least partial response
Evaluate Overall Survival in participants treated with Naïve HBI0101 CART | 24 Months after infusion
Evaluate Progression-Free Survival in participants treated with Naïve HBI0101 CART | 24 Months after infusion
Evaluate Duration of Response in participants treated with Naïve HBI0101 CART | 24 Months after infusion
Evaluate proportion of MRD negative subjects in participants treated with Naïve HBI0101 CART. | 24 Months after infusion
Evaluate persistence of Naïve HBI0101 CART in treated participants | 24 Months after infusion
  Quantification of Naïve HBI0101 CART in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah MO, Jerusalem, 9574869, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided